CLINICAL TRIAL: NCT02241499
Title: Palliative Short-course Hypofractionated Radiotherapy Followed by Chemotherapy in Adenocarcinoma of the Esophagus or Esophagogastric Junction Trial - a Phase II Clinical Trial Protocol.
Acronym: PALAESTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBG01
Record Dates: First submitted 2014-09-08; First posted 2014-09-16 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Adenocarcinoma of the Esophagus or Esophagogastric Junction
Keywords: Digestive System Diseases; Esophageal cancer; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Endoscopic response; Fluorouracil; Metabolic response; Oxaliplatin; Radiotherapy
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Digestive System Diseases; Esophageal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms | interventions — Radiotherapy; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy and chemotherapy (oxaliplatin and fluorouracil). (Experimental): Radiotherapy (5 x 4 Gy) will be given. After completion of radiotherapy, 4 cycles of chemotherapy will be administered, cycle length 14 days. Each patient will receive oxaliplatin as infusion at a dose of 85 mg/m2, followed by a bolus injection of fluorouracil at a dose of 400 mg/m2, and a long time infusion (44 hours) of fluorouracil at a dose of 2 400 mg/m2.
  Interventions: Radiation: Radiation therapy; Drug: Oxaliplatin and fluorouracil.

INTERVENTIONS:
Radiation: Radiation therapy — Radiotherapy at a dose of 4 Gy will be given to a total dose of 20 Gy, treatment duration 5 days.
Drug: Oxaliplatin and fluorouracil. — Oxaliplatin at a dose of 85 mg/m2 and will be given on day 1, infusion (44 hours) of fluorouracil will be given for 4 cycles, cycle length 14 days.

SUMMARY:
In this trial, patients with histologically proven adenocarcinoma of the esophagus or esophagogastric junction noneligible for surgery or chemoradiation with curative intent will be included. Primary objective is to determine the rate of improvement in dysphagia after palliative short course hypofractionated radiotherapy (5 x 4 Gy) followed by chemotherapy consisting of oxaliplatin and fluorouracil. The rate of improvement of dysphagia is evaluated by a 5 graded dysphagia score, and a positive change of at least 1 score is considered to be an improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven adenocarcinoma of the esophagus or esophagogastric junction noneligible for surgery or chemoradiation with curative intent
* Any T, N and M
* Age: 18 years or older
* WHO performance status ≤ 2
* Life expectancy > 3 months
* Dysphagia score > 0
* Adequate laboratory findings: hemoglobin > 90 g/L, absolute neutrophil count

  * 1.0 10 9/L, platelets ≥ 75 x 10 9/L, bilirubin ≤ 1.5 x upper limit of normal (ULN), alanine aminotransferase (ALAT) ≤ 5 x ULN, creatinine ≤ 1.5 x ULN
* Fertile men and women must use effective means of contraception
* Signed written informed concent
* The patient must be able to comply with the protocol

Exclusion Criteria:

* Prior treatment with self-expanding metal stent (SEMS), radiotherapy or chemotherapy for the present disease
* Clinically significant (i.e. active) cardiovascular disease e.g. myocardial infarction (≤ 6 months) unstable angina, New York Heart Association (NYHA) grade III-IV congestive heart failure
* Severe pulmonary disease e.g. pulmonary fibrosis
* Symptomatic peripheral neuropathy greater than grade 1 (CTCAE v. 4.0)
* Known hypersensitivity to any contents of the study drugs
* Pregnancy ( positive pregnancy test) and/or breast feeding
* Any other serious or uncontrolled illness which in the opinion of the investigator makes it undesirable for the patient to enter the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Improvement of dysphagia. | The grade of dysphagia is evaluated before start of treatment, 1-4 weeks after end of radiotherapy, then until local intervention or death, average of 12 months.
  The rate of improvement in dysphagia after palliative short course hypofractionated radiotherapy (5 x 4 Gy) followed by chemotherapy consisting of oxaliplatin and fluorouracil is evaluated by a 5 graded dysphagia score, and a positive change of at least 1 score is considered to be an approvement.

SECONDARY OUTCOMES:
Endoscopic response of the primary tumor. | Endoscopy will be performed before start of treatment, and within 4 weeks after end of radiotherapy.

OTHER OUTCOMES:
Metabolic response | Metabolic response will be evaluated before start of treatment, and within 4 weeks after end of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: David Borg, MD, Principal Investigator — Lund University Hospital, Department of Oncology
Locations (1):
- Lund University Hospital, Department of Oncology, Lund, Sweden